CLINICAL TRIAL: NCT04840186
Title: EXtended CriteriA Treatment for LIver Metastases and Heavy Tumour BURden
Acronym: EXCALIBUR3
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Lassen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 167434
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Liver Metastases; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: Multicentre RCT with two parallell arms. One with second line chemotherapy (standard care) and the other with second line chemotherapy + resection. We estimate an overall survival of 12 months in the standard care group. We aim to decide whether resections added to chemotherapy can increase this to 24 months. A two-sided parallel-group test of proportions to answer this with a power of 0.80 and an alpha of 0.15, will require 28 completed patients per group to show superiority for resections. Adding 11 % for a modified intention-to-treat analysis, we aim to randomise a total of 62 patients, i.e. 31 patients per group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2nd line chhemotherapy (Active Comparator): Patients in this arm will be receiving the standard care which is 2nd line chemotherapy. Type of chemotherapy determined by treating oncologist.
  Interventions: Drug: 2nd line chemotherapy
- 2nd line chemotherapy + resection (Active Comparator): Patients in this arm will be treated with liver resection and/or ablation at Oslo University Hospital followed by adjuvant 2nd line chemotherapy. Type of chemotherapy is determined by treating oncologist.
  Interventions: Procedure: Liver-resection or ablation; Drug: 2nd line chemotherapy

INTERVENTIONS:
Procedure: Liver-resection or ablation — Liver-resection of colorectal liver metastasis. Ablation can be used as adjunct to surgery.
  Arms: 2nd line chemotherapy + resection
Drug: 2nd line chemotherapy — 2nd line chemotherapy. Type of chemotherapy is determined by treating oncologist

SUMMARY:
Patients with multiple colorectal liver metastases that progress on 1st line chemotherapy have a very dismal prognosis, and their options are few. Resections are regularly performed although this is only supported by anecdotal evidence for this patient group. We want to assess whether resections actually confer benefit as compared to 2nd line chemotherapy alone, in a randomized controlled trial.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most frequent malignant disease in Norway (Cancer in Norway 2017). About 50% of the patients will have metastatic disease at the time of diagnosis or develop metastatic disease later on. Liver metastases are the most frequent presentation of metastatic disease. Liver resection is considered the only curative treatment option in CRC patients with liver metastases, however only about 20% of the patients are candidates for liver resection. The treatment option for the majority of the patients is palliative chemotherapy with a median overall survival from start of chemotherapy of about 2 years, and only 10-12 months from starting 2nd line chemotherapy.

While high-quality data (randomized trials) is wanting, it is generally accepted that the only curative treatment for colorectal liver metastases (CRLM) is surgery. Liver resections are generally well tolerated and safe 1, but some patients recur early and probably have no benefit from surgery, or even a net loss of quality-of-life (QoL). These are hard to identify beforehand, but patients with multiple tumours that progress on 1st line chemotherapy are at high risk of early recurrence following resection2, 3. These patients are in a grey zone: their metastases may be technically resectable, but the aggressive biology of their disease makes overall outcome of surgery highly uncertain. The decision to offer resection to some of these patients primarily results from want of better alternatives and from lack of sufficiently precise prognostication.

As resections are generally well tolerated and adequate prognostication is wanting, there is a tendency to offer resections to patients who have borderline resectable CRLM or who exhibit other non-favourable traits like large or multiple metastases, or progression on 1st line chemotherapy. Resections followed by early recurrence represent a net loss of quality-of-life and an unwanted expenditure for society. Exploring the optimal treatment modality for patients in this grey zone, i.e. with uncertain benefit from surgery, is important to provide optimal treatment for patients in a critical situation.

Palliative chemotherapy is in general the only treatment option for the vast majority of non-resectable patients. The expected median overall survival (OS) from start of first line chemotherapy is about 2 years and the 5 years OS is about 10%, although longer median OS has been obtained in selected patients with good performance status (ECOG 0-1), no (K)RAS or BRAF mutations and left-sided tumours 4-8. The OS from start of second line chemotherapy however is only 10-12 months 9. This places the prognosis for this group of cancer patients on par with those having pancreatic cancer.

This trial targets a group of patients that are not eligible for the Excalibur 1 and 2 trials but still have as dismal or even worse prognosis. They will - according to the inclusion criteria - have a large tumour burden and have shown progression on 1st line systemic chemotherapy treatment. Based on previous trials, only 30 % of this patient group are estimated to be alive after two years. These patients have today only one treatment modality available: 2nd line systemic chemotherapy. Response can, however, only be expected in a small minority.

With such a dismal outcome for these patients, almost any attempt to improve survival would be warranted and anecdotal evidence shows that some appear to benefit substantially. This may, however, be a result of biased selection and the benefit of surgery in this grey zone is unproven.

ELIGIBILITY:
Inclusion Criteria:

1. Verified adenocarcinoma in colon or rectum
2. Liver metastases that are technically resectable (ablation can be used as an adjunct) without PVE, HVE or ALPPS, but judged in need of further (next line) chemotherapy based on insufficient response to at least one line of chemotherapy. And either

   a. Six or more liver metastases, with extra-hepatic disease i. def: >3 pulmonary metastases/radiologically positive non-liver hilar lymph nodes. Or b. Ten or more liver metastases with at least one of the following negative prognostic signs: i. At least one lesion > 7 cm in diameter before chemotherapy ii. CEA > 100 following a full cycle of chemotherapy)?? iii. KRAS and/or BRAF mutant primary tumour. iv. Node positive primary tumour. Or c. Fifteen or more liver metastases
3. ECOG 0/2
4. Informed consent

Exclusion Criteria:

Any of the following criteria will exclude participation in the trial:

1. New liver metastases emerging during completed chemotherapy.

   a. These patients may be included if they undergo a complete cycle of next line chemotherapy without new liver metastases emerging.
2. Previous or current bone or CNS metastatic disease
3. Any other reason why, in the opinion of the investigators, the patient should not participate.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Median overall survival | 2years
  Primary endpoint is median survival after two years to see if the survival is different in the two groups.

SECONDARY OUTCOMES:
Quality of Life | EQ-5D-5L will be obtained at inclusion, week 6,12,18,24,36,48,60,72,84,96,108.
  Quality of life will analyzed by EuroQoL Group questionaire EQ-5D-5L
Progression free survival PFS | From inclusion to sign of progresion, tentatively less than 14months.
  Time from inclusion to sign of progression defined by the RECIST-criteria
Quality of life | EORTC QLQ-C30 will be obtained at inclusion, week 6,12,18,24,36,48,60,72,84,96,108.
  Quality of life will be analyzed by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Lassen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes